CLINICAL TRIAL: NCT04448054
Title: Imaging SARS-CoV-2 Involvement of Leptomeninges, Olfactory and Limbic Areas
Acronym: ICILOLA
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: 2020-A01216-33
Record Dates: First submitted 2020-06-23; First posted 2020-06-25 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Estimate, With the Contribution of Optimized MRI, the Prevalence of Neurological and Neurovascular Manifestations on Imaging in the Event of SARS-CoV-2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: MRI — Case 1: Routine care protocol not requiring injection
  * Realization of the non-injected MRI protocol adapted to the indication
  * + Addition of a 3D bFFE-Xd sequence (+ 2 min) The protocol will last the examination time usually provided by the current treatment according to the indication + 2 min of complementary sequence Case 2: Routine treatment protocol requiring an injection
  * Realization of the injected MRI protocol adapted to the indication
  * Before gadolinium injection:
  * Addition of a 3D bFFE-Xd sequence (+ 2 min) before injection
  * After gadolinium injection:
  * Option 1: if olfaction disorder, addition of DCE perfusion sequence (T1-WI) which will be the 1st post injection sequence (+ 4 min 30)
  * FABIR 0.9 3D sequence (+ 4 min)
  * 3D sequence T1 TSE 0.7 (+ 2 min 30)
  * FLAIR HR coronal sequence (+ 3 min 30)
  * Option 2: if hearing / balance disorder, adding 3D FLAIR "labyrinth" sequence (+ 6min) which will be the 1st post injection sequence

SUMMARY:
When patients arrive in the waiting room of the MRI department, patients will be given the briefing note explaining the purpose of the study and how it is going. During the consultation, the radiologist will check the inclusion and non-inclusion criteria, and will take the time to answer all of the patient's questions about the study (or his family member by telephone if the patient does not is not in a condition to give its consent).

The MRI examination will be performed on a 3T multi-parametric MRI. If the neurological disorder presented by the patient does not require an injection as part of routine care, only a high resolution 3D T2 sequence on the nasosinus cavities and the olfactory tract, called bFFE-Xd for approximately 2 min.

If the neurological disorder presented by the patient requires an injection as part of current care, the examination will be completed with the nasosinus and olfactory 3D bFFE-Xd sequence, and the following additional sequences performed after post injection: a

* 3D FABIR 0.9 sequence covering the brain, dedicated to exploring the subarachnoid spaces;
* a 3D T1 TSE 0.7 sequence covering the brain looking for meningeal or encephalic contrast enhancement,
* FLAIR HR coronal sequence (high resolution) exploring the limbic system.
* Optional: a 3D FLAIR "labyrinth" sequence in the event of hearing / balance problems; a DCE infusion sequence (T1-WI) on the olfactory tract if olfactory disorder, which will be the first sequence made at the time of injection.

ELIGIBILITY:
Inclusion Criteria:

Patient> 18 years old Express consent to participate in the study Affiliate or beneficiary of a social security scheme Patient with suspected SARS-CoV-2 infection in an epidemic context, confirmed or not by PCR, or close contact with a case confirmed by PCR, typical chest scanner (non-systematized frosted glass areas predominantly sub-pleural, and at a later stage of alveolar condensation without excavations, nodules or masses) or positive serology; Patient to benefit from a brain MRI for an indication within the scope of care

Exclusion Criteria:

Patient benefiting from a legal protection measure Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient diagnosed with SARS-CoV-2, who should benefit from a brain MRI as part of care for an acute / chronic neurological disorder.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Percentage of patients included with at least one sign of neuromeningeal, neurosensory or neurovascular involvement on MRI imaging with the specific sequences used. | baseline
  percentage

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation A De Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No